CLINICAL TRIAL: NCT01578655
Title: A Randomized Phase 3 Study Comparing Cabazitaxel/Prednisone in Combination With Custirsen (OGX-011) to Cabazitaxel/Prednisone for Second-Line Chemotherapy in Men With Metastatic Castrate Resistant Prostate Cancer (AFFINITY)
Brief Title: Comparison of Cabazitaxel/Prednisone Alone or in Combination With Custirsen for 2nd Line Chemotherapy in Prostate Cancer
Acronym: AFFINITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OGX-011-12
Record Dates: First submitted 2012-04-09; First posted 2012-04-17 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: custirsen sodium; prostate cancer; metastatic castrate resistant prostate cancer; overall survival
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; Prednisone; OGX-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabazitaxel plus Custirsen (Experimental): cabazitaxel, prednisone, and custirsen sodium
  Interventions: Drug: cabazitaxel; Drug: prednisone; Drug: custirsen sodium
- Cabazitaxel (Active Comparator): cabazitaxel and prednisone
  Interventions: Drug: cabazitaxel; Drug: prednisone

INTERVENTIONS:
Drug: cabazitaxel — Cabazitaxel (25mg/m² IV) is administered on day 1 of each 21-day cycle until disease progression, unacceptable toxicity, or completion of 10 cycles
Drug: prednisone — Prednisone (10 mg PO) is administered daily until disease progression, unacceptable toxicity, or completion of 10 cycles
Drug: custirsen sodium — Custirsen is administered as 3 loading doses (640 mg IV each) within 9 days, followed by weekly custirsen (640 mg IV) during each 21-day cycle until disease progression, unacceptable toxicity, or completion of 10 cycles
  Other Names: OGX-011; TV-1011
  Arms: Cabazitaxel plus Custirsen

SUMMARY:
This Phase 3 study has been designed to confirm that adding custirsen to cabazitaxel/prednisone treatment can slow tumor progression and enhance survival outcomes compared to standard cabazitaxel/prednisone treatment in men with metastatic castrate resistant prostate cancer (CRPC). This will be a randomized, open-label, multicenter, international trial. Treatment will consist of cabazitaxel/prednisone/custirsen vs. cabazitaxel/prednisone. A total of approximately 630 patients will be randomized with equal probability to the two arms.

DETAILED DESCRIPTION:
Until recently, options for second-line chemotherapy in CRPC have included docetaxel retreatment, mitoxantrone, or other chemotherapies, without proven clinical benefit. In 2010, a Phase 3 second-line chemotherapy trial (TROPIC) showed a survival advantage for cabazitaxel, a semi-synthetic taxane selected to overcome the emergence of taxane resistance, when compared to mitoxantrone.

Clusterin is a stress-activated cytoprotective chaperone up-regulated by a variety of anti-cancer therapies that confers treatment resistance when over-expressed. Inhibition of clusterin expression using custirsen has been shown to enhance tumor cell death following treatment with chemotherapy.

The clinical activity of custirsen in combination with the taxane docetaxel has been shown in two Phase 2 studies. Given the results observed using a taxane as either first-line or second-line chemotherapy in CRPC, combination with custirsen may decrease taxane resistance and enhance the survival benefit of taxane therapy. Thus, a combination of custirsen with cabazitaxel may further enhance survival in second-line taxane chemotherapy for CRPC.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of adenocarcinoma of the prostate
* Metastatic disease on chest, abdominal, or pelvic CT scan and/or bone scan
* Previous first-line treatment for CRPC with a docetaxel-containing regimen
* Current progressive disease
* Increasing serum PSA level (for patients who progress based only on increasing serum PSA level, a minimum starting value of 5.0 ng/mL is required)
* Baseline laboratory values as defined
* Willing to continue primary androgen suppression with gonadotropin-releasing hormone (GnRH) analogues (unless treated with bilateral orchiectomy)
* Karnofsky score ≥70%
* At least 21 days have passed since completing radiotherapy
* At least 21 days have passed since receiving any investigational agent at the time of randomization
* At least 21 days have passed since major surgery
* Recovered from any docetaxel therapy-related neuropathy to ≤grade 1 at the time of randomization
* Recovered from all therapy related toxicity to ≤grade 2 (except alopecia, anemia, and any signs or symptoms of androgen deprivation therapy) at the time of randomization
* Able to tolerate a starting dose of 25 mg/m² cabazitaxel
* Willing to not add, delete, or change current bisphosphonate or denosumab usage
* Able to tolerate oral prednisone at 10 mg per day
* Competent to provide written informed consent

Exclusion Criteria:

* Received any other cytotoxic chemotherapy beyond the first-line docetaxel-containing regimen as treatment for prostate cancer
* Received prior radioisotope with strontium 89 or samarium 153
* Received any cycling, intermittent, or continuous hormonal treatment within 21 days prior to randomization with the exception of the continuous GnRH analogues (prior treatment with abiraterone or MDV3100 is allowed as long as 21 days have passed since last dose)
* Participated in a prior Phase 3 clinical study evaluating custirsen regardless of study arm assignment
* Requiring ongoing treatment during the study with medications known to be either strong CYP3A inhibitors or strong CYP3A inducers
* History of or current documented brain metastasis or carcinomatous meningitis, treated or untreated
* Current symptomatic cord compression requiring surgery or radiation therapy
* Active second malignancy (except non melanomatous skin or superficial bladder cancer) defined in general as requiring anticancer therapy or at high risk of recurrence during the study
* Uncontrolled medical condition or significant concurrent illness that in the opinion of the Investigator would preclude protocol therapy
* Known severe hypersensitivity to taxanes or polysorbate 80-containing drugs
* Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2012-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Survival in the intent-to-treat population | 3.4 years
  To determine whether the survival for patients randomized to the investigational arm (cabazitaxel/prednisone plus custirsen) is consistent with longer survival as compared to patients randomized to the control arm (cabazitaxel/prednisone).
Survival in the poor-prognosis patient population | 2.7 years
  To determine whether the survival for patients randomized to the investigational arm (cabazitaxel/prednisone plus custirsen) and identified as having poor prognosis is consistent with longer survival as compared to patients randomized to the control arm (cabazitaxel/prednisone) and identified as having poor prognosis.

SECONDARY OUTCOMES:
Progression-free survival at Day 140 | From randomization to Day 125 to Day 155
  To compare the arms with respect to the proportion of patients having a milestone Day 140 status of Alive Without Event (within the window of Day 125-155 post-randomization). An event is defined as disease progression or death on or before Day 140.

CONTACTS AND LOCATIONS:
Overall Officials: Thomasz Beer, MD, Principal Investigator — Oregon Health & Science University, Portland, Oregon; Karim Fazazi, MD, Principal Investigator — Gustave Roussy Cancer Institute, University of Paris, France; Sebastien Hotte, MD, Principal Investigator — Juravinski Cancer Centre, Hamilton, Ontario, Canada
Locations (94):
- United States (35):
  - Prostate Oncology Specialists, Marina del Rey, California
  - University of California Davis Medical Center, Sacramento, California
  - Sharp Health Care, San Diego, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Rocky Mountain Cancer Center, Boulder, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital at Yale New Haven Hospital, New Haven, Connecticut
  - The Center for Hematology-Oncology, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, Inverness, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Georgia Cancer Specialists, P.C., Marietta, Georgia
  - Cancer Center of Kansas, Wichita, Kansas
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Urology Cancer Center and GU Research Network, Omaha, Nebraska
  - Monter Cancer Center, Lake Success, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Albert Einstein Medical Center, The Bronx, New York
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Oncology Hematology Care, Inc., Blue Ash, Ohio
  - The Mark H. Zangmeister Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology, PA, Dallas, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
- Australia (11):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St George Public Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Haematology and Oncology Clinics of Australia, Brisbane, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Epworth Healthcare, Richmond, Victoria
- Canada (8):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - R. S. McLaughlin Durham Regional Cancer Center at Lakeridge Health Oshawa, Oshawa, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHUM-Hospital Notre-Dame, Montreal, Quebec
- Czechia (4):
  - Krajská nemocnice Liberec a.s., Liberec, Liberec
  - Krajská nemo. T.Bati, a. s., Zlín, Severomoravsky Kraj
  - Fakultni nemo Hradec Králové, Hradec Králové
  - University Hospital Olomouc, Olomouc
- France (10):
  - Centre Léon Bérard, Lyon Cédex 08, Auvergne-Rhône-Alpes
  - Centre François Baclesse, Caen, Basse-Normandie
  - Institut Jean-Godinot, Reims, Champagne-Ardenne
  - Institut Paoli Calmettes, Marseille, Marseille
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Poitiers Hôpital de la Milétrie, Poitiers, Poitou-Charentes
  - Centre Antoine Lacassagne, Nice, Provence-Alpes-Côte d'Azur Region
  - Hôpital Saint Louis, Paris, Île-de-France Region
  - Institut Curie, Paris, Île-de-France Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Hungary (5):
  - Pándy Kálmán Megyei Kórház, Gyula, Bekes County
  - Borsod Abaúj Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc, Borsod-Abauj Zemplen county
  - Országos Onkológiai Intézet, Budapest, Budapest
  - Semmelweis Egyetem Általános Orvostudományi Kar, Budapest, Budapest
  - Szegedi Tudományegyetem, Onkoterápiás Klinika, Szeged, Csongrád megye
- Russia (12):
  - Ivanovo Reg Oncology Centre, Ivanovo, Ivanovo Oblast
  - Cancer Research Center na NN Blokhin, Moscow, Moscow
  - Hertzen Rsrch Inst of Oncology, Moscow, Moscow
  - Sverdlovsk Reg Clin Hosp#1, Yekaterinburg, Ural
  - Volgograd Regional Oncological Dispensary, Volzhsky, Volgograd Oblast
  - S Inst Hlth Altay Reg Onc Disp, Barnaul
  - Russian Research Center of Radiology, Moscow
  - Urology Research Institute, Moscow
  - State Healthcare Inst Omsk Reg, Omsk
  - Petrov Research Oncology Institute, Saint Petersburg
  - Saint Petersburg City Oncological Dispensary, Saint Petersburg
  - Stavropol Reg Oncology Ctr, Stavropol
- United Kingdom (9):
  - Cancer Research UK, Birmingham, England
  - Addenbrookes Hospital Cambridge, Cambridge, England
  - U of Surrey Post Grad Med, Guildford, England
  - Christie Hospital NHS Foundation Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Foundation Trust, Metropolitan Borough of Wirral, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - The Royal Marsden Hospital, Surrey, England
  - Musgrove Park Hospital, Taunton, England
  - Beatson Cancer Centre, Glasgow, Glasgow, Scotland

REFERENCES:
- [Background] Saad F, Hotte S, North S, Eigl B, Chi K, Czaykowski P, Wood L, Pollak M, Berry S, Lattouf JB, Mukherjee SD, Gleave M, Winquist E; Canadian Uro-Oncology Group. Randomized phase II trial of Custirsen (OGX-011) in combination with docetaxel or mitoxantrone as second-line therapy in patients with metastatic castrate-resistant prostate cancer progressing after first-line docetaxel: CUOG trial P-06c. Clin Cancer Res. 2011 Sep 1;17(17):5765-73. doi: 10.1158/1078-0432.CCR-11-0859. Epub 2011 Jul 25. PMID 21788353
- [Background] Chi KN, Hotte SJ, Yu EY, Tu D, Eigl BJ, Tannock I, Saad F, North S, Powers J, Gleave ME, Eisenhauer EA. Randomized phase II study of docetaxel and prednisone with or without OGX-011 in patients with metastatic castration-resistant prostate cancer. J Clin Oncol. 2010 Sep 20;28(27):4247-54. doi: 10.1200/JCO.2009.26.8771. Epub 2010 Aug 23. PMID 20733135
- [Derived] Beer TM, Hotte SJ, Saad F, Alekseev B, Matveev V, Flechon A, Gravis G, Joly F, Chi KN, Malik Z, Blumenstein B, Stewart PS, Jacobs CA, Fizazi K. Custirsen (OGX-011) combined with cabazitaxel and prednisone versus cabazitaxel and prednisone alone in patients with metastatic castration-resistant prostate cancer previously treated with docetaxel (AFFINITY): a randomised, open-label, international, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1532-1542. doi: 10.1016/S1470-2045(17)30605-8. Epub 2017 Oct 9. PMID 29033099